CLINICAL TRIAL: NCT01979783
Title: Correlation Between Electromyography and Thickness Change of the Trunk Muscles in Subjects With Low Back Pain
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Olivera Djordjevic, medical doctor, University of Belgrade
Other Study IDs: EMGUS
Record Dates: First submitted 2013-10-28; First posted 2013-11-08 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-11

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day

GROUPS / COHORTS (2):
- LBP: group of subjects with low back pain
- nonLBP: group without low back pain

SUMMARY:
Transversus abdominis (TrA) and lumbar multifidus (LM) muscle have been proposed to play key role in stability of the lumbosacral spine. The muscles' functional and/or structural deficits have been linked to the low back pain (LBP) syndrome. Evaluation of the transversus abdominis and lumbar multifidus muscles' function in clinical practice is scarce and not well defined due to number of reasons. Surface electromyography of TrA and LM muscles, as a method of examining muscles function, is not involved in clinical routine. Rehabilitative Ultrasound Imaging (RUSI) of the TrA and LM, apart from providing information about their morphology, could be helpful in assessing their function. Since concentric muscle contraction results in the shortening and thickening of the muscle, evaluation of the potential association between muscle's morphometry, assessed by the ultrasound, and electromyography, may be of potential clinical interest. However, this potential relationship is context-dependant. Our aim was to establish the difference in the thickness change of the TrA and LM muscle during activation in subjects with and without low back pain, and to establish the possible correlation between electromyography and the thickness change of these muscles assessed by ultrasound in both groups of subjects.

ELIGIBILITY:
Inclusion Criteria:

Low back pain, with or without radiculopathy, that lasted for at least 12 weeks, caused by prolapsed intervertebral disc (PID), confirmed by magnetic resonance imaging (MRI)

Exclusion Criteria:

The exclusion criteria for all participants were pregnancy,diabetes mellitus,corticosteroids administrated in one months or less prior to enrollment, spinal fractures, surgery, infectious diseases, tumors, spina bifida, advanced forms of spinal deformity, hip diseases, and neuromuscular disorders. Additional exclusion criteria for LBP participants were self-reported pain levels of less than 3 on the Visual Analog Scale to account for patients commonly encountered in clinical practice, and inability to remain in prone and supine hook-lying positions for 10 minutes each in order to ensure compliance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: tertiary care clinic
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
thickness of the lumbar multifidus and transversus abdominis muscle | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic for Rehabilitation Dr Mirsoslav Zotovic Faculty of Medicine University of Belgrade, Belgrade, Serbia

REFERENCES:
- [Derived] Djordjevic O, Konstantinovic L, Miljkovic N, Bijelic G. Relationship Between Electromyographic Signal Amplitude and Thickness Change of the Trunk Muscles in Patients With and Without Low Back Pain. Clin J Pain. 2015 Oct;31(10):893-902. doi: 10.1097/AJP.0000000000000179. PMID 25380224